CLINICAL TRIAL: NCT00263692
Title: Open, Randomized, Phase II, Clinical Trial to Compare the Immunogenicity and Safety of a Booster Dose of GSK Biologicals' DTaP-IPV Vaccine (Infanrix®-IPV) Co-administered With a Booster Dose of Merck and Company's M-M-R®II, to That of Separate Injections of GSK Biologicals' DTaP Vaccine (Infanrix®), Aventis Pasteur's IPV (IPOL®) and M-M-R®II Administered as Booster Doses to Healthy Children 4 to 6 Years of Age.
Brief Title: Comparison of GSK Biologicals' DTaP-IPV Candidate Vaccine to DTaP and IPV Separately Administered Vaccines in Terms of Immune Response and Safety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 213503/047
Record Dates: First submitted 2005-12-08; First posted 2005-12-09 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Diphtheria; Acellular Pertussis; Tetanus
MeSH Terms: conditions — Diphtheria; Tetanus | interventions — Tetanus Toxoid

INTERVENTIONS:
Biological: Prophylaxis: Diphtheria, tetanus, pertussis, poliovirus type 1, type 2 and type 3

SUMMARY:
The aims of this study are to compare the immunogenicity and safety of the GSK Biologicals' combined DTaP-IPV vaccine with separate administration of DTaP and IPV vaccines, when administered as a fifth dose of acellular pertussis vaccine to children aged 4 to 6 years when co-administered with MMR vaccine in subjects who had previously received four doses of Infanrix, three doses of poliovirus-containing vaccine and MMR vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children between and including 4 and 6 years of age.
* Previously received 4 doses of GSK Biologicals' DTaP, 3 doses of IPV vaccine and 1 dose of measles, mumps, and rubella vaccine.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccines within 30 days preceding the administration of study vaccines, or planned use during the study period.
* Chronic administration or planned administration of immunosuppressants or other immune modifying drugs within six months prior to study vaccination or planned administration during the study period
* Administration of immunoglobulins and/or blood products within 3 months prior to vaccination.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 401 (Actual)
Dates: Start 2002-11; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Immunogenicity after vaccination.

SECONDARY OUTCOMES:
Immunogenicity and safety after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- United States (15):
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Ruston, Louisiana
  - GSK Investigational Site, Berlin, New Jersey
  - GSK Investigational Site, Whitehouse Station, New Jersey
  - GSK Investigational Site, Endwell, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Mechanicsville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Black S, Friedland LR, Schuind A, Howe B; GlaxoSmithKline DTaP-IPV Vaccine Study Group. Immunogenicity and safety of a combined DTaP-IPV vaccine compared with separate DTaP and IPV vaccines when administered as pre-school booster doses with a second dose of MMR vaccine to healthy children aged 4-6 years. Vaccine. 2006 Aug 28;24(35-36):6163-71. doi: 10.1016/j.vaccine.2006.04.001. Epub 2006 Apr 21. PMID 16759769
- [Background] Weston WM, Klein NP. Kinrix: a new combination DTaP-IPV vaccine for children aged 4-6 years. Expert Rev Vaccines. 2008 Nov;7(9):1309-20. doi: 10.1586/14760584.7.9.1309. PMID 18980534
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 213503/047 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 213503/047 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 213503/047 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 213503/047 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 213503/047 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 213503/047 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register